CLINICAL TRIAL: NCT05958498
Title: Consequence of Injectable Platelets Rich Fibrin Versus Microosteopeforationon Root Resorption During Orthodontic Intrusion of Incisor Teeth: A Comparative Clinical Study
Brief Title: Consequence of Injectable Platelets Rich Fibrin Versus Microosteopeforation on Root Resorption During Orthodontic Intrusion of Incisor Teeth
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Al-Azhar University (Other)
Responsible Party: Principal Investigator, farouk ahmed hussein, Principal Investigator, Al-Azhar University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 922/91
Record Dates: First submitted 2023-07-15; First posted 2023-07-24 (Actual); Last update posted 2023-07-24 (Actual); Status verified 2023-07

CONDITIONS: Compare the Effect of Injectable Platelets Rich Fibrin and Micro-osteoperforations on Root Resorption During Orthodontic Intrusion of Incisors

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group I (Active Comparator): who will receive intrusive arches after leveling and alignment assisted with i-PRF according to standardized protocol
  Interventions: Combination Product: injectable platelet rich fibrin and microosteoperforation
- Group II (Active Comparator): Will includes 9 patients who will receive intrusive utility arches after leveling and alignment assisted with (MOPs) according to standardized protocol.
  Interventions: Combination Product: injectable platelet rich fibrin and microosteoperforation

INTERVENTIONS:
Combination Product: injectable platelet rich fibrin and microosteoperforation — i-PRF which second product of blood versus mops which is surgical procedure

SUMMARY:
Consequence of injectable platelets rich fibrin versus microosteopeforation on root resorption during orthodontic intrusion of incisor teeth

DETAILED DESCRIPTION:
Consequence of injectable platelets rich fibrin versus microosteopeforation on root resorption during orthodontic intrusion of incisor teeth: A comparative clinical study

ELIGIBILITY:
Inclusion Criteria:

* 1. Patients with age range between 12-16 years. 2. Overbite > 40% indicated for maxillary intrusion. 3. Mild to moderate crowding of upper incisors. 4. All permanent teeth erupted (excluding 3rd molars). 5. No previous orthodontic treatment. 6. Good oral hygiene with no previous periodontal surgery.

Exclusion Criteria:

1. - Transverse and/or vertical skeletal dysplasia or craniofacial malformation. 2. Retained primary or missing permanent teeth in the maxillary anterior area, and any kind of tooth/root shape anomaly.

3. Patients with root resorption, impacted canines, or dental anomalies. 4. Poor oral hygiene 5. Present or history of periodontal diseases. 6. Systemic diseases or regular use of medications that could interfere with orthodontic tooth movement.

7. History of trauma affecting the maxillary incisors. 8. Endodontically treated upper anterior teeth.

Ages: 15 Years to 22 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 18 (Estimated)
Dates: Start 2023-12 (Estimated); Primary Completion 2024-06 (Estimated); Study Completion 2024-08 (Estimated)

PRIMARY OUTCOMES:
to compare the effect of injectable platelets rich fibrin and micro-osteoperforations on root resorption during orthodontic intrusion of incisors. | post interventionalal at 6months
  amount of root resorption

CONTACTS AND LOCATIONS:
Locations (1):
- AlAzhar university, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Zeitounlouian TS, Zeno KG, Brad BA, Haddad RA. Three-dimensional evaluation of the effects of injectable platelet rich fibrin (i-PRF) on alveolar bone and root length during orthodontic treatment: a randomized split mouth trial. BMC Oral Health. 2021 Mar 2;21(1):92. doi: 10.1186/s12903-021-01456-9. PMID 33653326
- [Background] Dos Santos CCO, Mecenas P, de Castro Aragon MLS, Normando D. Effects of micro-osteoperforations performed with Propel system on tooth movement, pain/quality of life, anchorage loss, and root resorption: a systematic review and meta-analysis. Prog Orthod. 2020 Jul 27;21(1):27. doi: 10.1186/s40510-020-00326-4. PMID 32715352